CLINICAL TRIAL: NCT02474550
Title: Multicenter Prospective Registry Study of Diffuse Large B Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Seong Hyun Jeong, Associate, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-14-254
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diffuse Large B Cell Lymphoma; Neutropenia, Febrile
Keywords: diffuse large b cell lymphoma; peg-filgrastim; febrile neutropenia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CISL 14-03: * Patients who were newly diagnosed with Diffuse Large B cell Lymphoma (DLBCL).
  * Aged 19 or more
  * Treated with R-CHOP therapy

SUMMARY:
This study was designed to review clincal outcomes of Diffuse Large B Cell Lymphoma (DLBCL) treated with R-CHOP chemotherapy in the era of pegylated-filgrastim. The investigators will prospectively collect clinical data and treatment outcome of patients with DLBCL who use prophylactic pegylated-filgrastim.

DETAILED DESCRIPTION:
* Newly diagnosed DLBCL patients treated with R-CHOP chemotherapy
* Prphylactic peg-filgrastim on the day after chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* 19 or older
* newly diagnosed with DLBCL
* R-CHOP chemotherapy
* offer informed consent

Exclusion Criteria:

* other subtype of NHL
* concomitant other cancer
* previous chemotherapy or radiotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with DLBCL in Korea
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
incidence of febrile neutropenia | within 30 days

SECONDARY OUTCOMES:
incidence of chemotherapy-related adverse events other than febrile neutropenia | 4 weeks after completion of chemotherapy
Overall survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hyun Jeong, M.D, Principal Investigator — Ajou University School of Medicine
Locations (24):
- South Korea (24):
  - Ajou Universtiy School of Medicine, Suwon, Kyeonggi
  - Soon Chun Yang University Hospital Bucheon, Bucheon-si
  - Busan Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung Univerisity Dongsan Medical Center, Daegu
  - Yeungnam University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon University Gill Hospital, Incheon
  - Chonbuk Nationa University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Asan Medical Center, Seoul
  - Choong Ang University Hopspital, Seoul
  - Hallym University Sacred Heart Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Korea Institute of Radiological & Medical Science, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No